CLINICAL TRIAL: NCT06974435
Title: Efficacy of Interval Training and Low-Frequency Pulsed Electromagnetic Field Therapy on Improving Cardiovascular Disease Risk and Lower Extremity Function in Diabetic Elderly: Randomized Controlled Trial
Brief Title: Interval Training and Electromagnetic Therapy on Cardiovascular Disease Risk in Diabetic Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umm Al-Qura University (Other)
Responsible Party: Principal Investigator, Ashraf Abdelaal, Associate Professor, Umm Al-Qura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HAPO-02-K-012-2022-03-997
Record Dates: First submitted 2025-05-07; First posted 2025-05-15 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Cardiovascular Disease Risk Reduction; Diabetes; Lower Extremity Dysfunction
Keywords: Cardiovascular disease risk; Exercise; Magnetic Therapy; Lower Limb Function; Diabetes
MeSH Terms: conditions — Diabetes Mellitus; Motor Activity | interventions — Magnetic Field Therapy; Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group-A (interval training and electromagnetic therapy group; n=25) (Experimental): Group A: received moderate intensity interval training in addition to low-frequency pulsed electromagnetic field therapy. The treatment program was in the form of twice-weekly sessions for 8 weeks, in addition to medical treatment.
  Interventions: Behavioral: Interval training and electromagnetic therapy
- Group-B (electromagnetic therapy group; n=25) (Experimental): Group B: received low-frequency pulsed electromagnetic field therapy only. The treatment program was in the form of twice-weekly sessions for 8 weeks, in addition to medical treatment.
  Interventions: Behavioral: Electromagnetic therapy
- Group-C (interval training group; n=25) (Experimental): Group C: received moderate intensity interval training. The treatment program was in the form of twice-weekly sessions for 8 weeks, in addition to medical treatment.
  Interventions: Behavioral: Interval exercise training
- Control group (Group; No-intervention group) (Other): Control group (Group; No-intervention group): received only the medical treatment.
  Interventions: Other: Control group (No intervention group)

INTERVENTIONS:
Behavioral: Interval training and electromagnetic therapy — Combined application of moderate intensity interval training and low frequency pulsed electromagnetic field therapy, in addition to pharmacotherapy.
  Arms: Group-A (interval training and electromagnetic therapy group; n=25)
Behavioral: Interval exercise training — Application of moderate intensity interval training, in addition to pharmacotherapy.
  Arms: Group-C (interval training group; n=25)
Behavioral: Electromagnetic therapy — Application of low-frequency pulsed electromagnetic field therapy, in addition to pharmacotherapy.
  Arms: Group-B (electromagnetic therapy group; n=25)
Other: Control group (No intervention group) — Only Pharmacotherapy.
  Arms: Control group (Group; No-intervention group)

SUMMARY:
Aims: To evaluate the combined effect of moderate intensity interval training and low frequency pulsed electromagnetic field therapy on cardiovascular disease risk and lower extremity functioning in the elderly with type 2 diabetes mellitus.

Methods: One hundred patients with type 2 diabetes mellitus were randomly allocated into four groups: group A (received moderate intensity interval training+low frequency pulsed electromagnetic field therapy; n=25), group-B (received low frequency pulsed electromagnetic field therapy only; n=25), group C (received moderate intensity interval training only; n=25), and (control group; no intervention; n=25). Treatment programs for groups A, B, and C were in the form of twice-weekly sessions for 8 weeks. Variables were evaluated at the beginning and the end of the study. The cardiovascular disease risk (evaluated using the Atherosclerotic Cardiovascular Disease risk estimator plus tool, Framingham Cardiovascular Disease risk estimation tool, and the mean arterial pressure methods). Lower extremity functioning was evaluated using the Short Physical Performance Battery. Within and between-subjects statistical comparisons were performed to test the hypothesis (to test whether the combined application of moderate intensity interval training+low frequency pulsed electromagnetic field therapy is effective in improving the cardiovascular disease risk and lower limbs functional status in ethe lderly with type 2 diabetes mellitus), A P-value of <0.05 was considered significant.

DETAILED DESCRIPTION:
Diabetes mellitus is a continuously growing epidemic all over the world. The continuously increasing number of patients with diabetes mellitus and its complications is a serious challenge to patients and health care providers. Cardiovascular disease is the primary cause of death in patients with diabetes mellitus worldwide. The presence of diabetes mellitus in addition to getting older magnifies the cardiovascular disease risk and predisposes to its occurrence at an earlier age. The prevalence of different cardiovascular disease types within patients with diabetes reached 18 % in Saudi Arabia.

The Lower limb diabetes-related complications are common and usually associated with increased morbidity and mortality. Diabetes mellitus contributes significantly to the development of peripheral vascular disorders, ischemia, and even amputation. A strong correlation exists between Diabetes mellitus and cardiovascular disease, about 44% and 52% of deaths in patients with type 1 and type 2 diabetes mellitus, respectively, are due to cardiovascular disease. Diabetes mellitus magnifies the chance of dying from cardiovascular disorders by two to four times in patients with diabetes compared to those without diabetes. This fact highlights the importance of introducing cardiovascular disease risk-reduction strategies in the management programs.

Furthermore, cardiovascular disease risk is proportionally increased and correlated with the hyperglycemia status even before diabetes diagnosis. The existence of other factors, such as hypertension, dyslipidemia, and obesity, accelerates the development of cardiovascular disease in patients with diabetes. So, early identification and management of cardiovascular disease risk is a major concern during diabetes mellitus management. Diabetes mellitus is tightly correlated as a causative agent to peripheral circulatory disturbances, limb ischemia, and even amputation. Early and proper management of the diabetes-related lower limb abnormalities is crucial for minimizing complications and dysfunction.

Moderate to high-intensity interval training is commonly included in the management programs for patients with type 2 diabetes mellitus. Studies demonstrated favorable effects of exercise training on cardiovascular and metabolic parameters in patients with diabetes mellitus. Physical training can improve cardiopulmonary and metabolic variables that, in turn, can ameliorate complications' progression and improve disease prognosis.

Engagement in regular physical training can significantly reduce the cardiovascular disease risk. An increase of weekly activity hours by 11.25 metabolic equivalents can reduce cardiovascular disease mortality by 23%. Increased physical activity has a positive impact on cardiovascular, musculoskeletal, metabolic, and psychosocial function in patients with DM, resulting in a lower mortality rate.

Low-frequency pulsed electromagnetic field therapy has beneficial and prognostic impacts on metabolic profile in patients with type 2 diabetes mellitus due to its favorable, vasoactive, neuro-stimulatory, and analgesic effects. Studies clarified favorable effects of therapeutic pulsed electromagnetic field application on different musculoskeletal, cardiovascular, and metabolic parameters in patients with type 2 diabetes mellitus. A Recent study demonstrated significant effects of cross-over application of the electromagnetic field therapy and interval exercise training on the balance and peripheral vascular status in patients with diabetes mellitus.

To our knowledge and recent literature, no study has investigated the effects of combined application of both interval training and low-frequency pulsed electromagnetic field therapy on cardiovascular disease risk and lower extremity function in older adults with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary older adult (65-75 years old).
* Diagnosed with type 2 diabetes mellitus.
* Glycosylated hemoglobin ≥ 6.5%.
* Receiving oral anti-diabetic medications only.
* Cognitively competent and able to understand and follow instructions.

Exclusion Criteria:

* Patients younger than 65 or older than 75.
* Diagnosed with type 1 diabetes.
* Included in an active exercise training or physiotherapy program within the last 6 months.
* With serious cardiac insults as myocardial infarction, lower limbs metal implants (internal fixation).

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-03-07 (Actual); Study Completion 2025-04-06 (Actual)

PRIMARY OUTCOMES:
Change in the cardiovascular disease risk at 8-week. | From enrollment to the end of treatment at 8 weeks.
  The cardiovascular disease risk was evaluated using the Atherosclerotic Cardiovascular Disease risk estimator plus tool, the Framingham Cardiovascular Disease risk estimation tool, and the mean arterial pressure methods.
Change in the lower extremity functioning at 8-week. | From enrollment to the end of treatment at 8 weeks.
  Lower extremity functioning was evaluated using the Short Physical Performance Battery.

CONTACTS AND LOCATIONS:
Overall Officials: ASHRAF AM ABDELAAL, Ph.D., Principal Investigator — Associate Professor
Locations (1):
- Umm Al-Qura University, Mecca, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
For privacy reasons, data can not be exposed until results' publication. Data summary will be confidentially provided upon request under limited situations.